CLINICAL TRIAL: NCT02089789
Title: Clinical and Basic Investigations Into Known and Suspected Congenital Disorders of Glycosylation and Deglycosylation
Brief Title: Clinical and Basic Investigations Into Known and Suspected Congenital Disorders of Glycosylation
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140071; 14-HG-0071
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-28

CONDITIONS: Congenital Disorders of Glycosylation
Keywords: Thrombosis; Intellectual Disability; Hypotonia; Hypoglycemia; Hypothyroidism; Natural History
MeSH Terms: conditions — Congenital Disorders of Glycosylation; Thrombosis; Intellectual Disability; Muscle Hypotonia; Hypoglycemia; Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CDG: Patients with a suspected CDG based on biochemical tests or a confirmed CDG based on enzymatic or molecular tests will be eligible to enroll in this protocol

SUMMARY:
Background:

- Proteins, fats, and other molecules are the body s building blocks. Many of these molecules must have sugars, or chains of sugars, attached to work properly. People with congenital disorders of glycosylation (CDGs) cannot attach these sugars or sugar chains properly. A child or adult with a CDG can have symptoms in different parts of the body, including brain, nerves, muscles, liver, and immune system. Researchers want to learn more about these diseases to understand better what is causing the problems.

Objective:

- To learn more about CDGs.

Eligibility:

- People 1 month to 2 years old may be seen as outpatients or by telehealth. Patients 2-80 years with CDG or suspected to have a CDG may be seen under this protocol as inpatients, outpatients or by teleheath.

Design:

* CDG participants may be seen as inpatients, outpatients or by teleheath. Inpatient stays may last 2-5 days.
* They will have:-Medical history and physical exam. They will answer questions about their CDG.
* Blood taken several times. Their skin will be numbed, then a needle will take blood from an arm vein.
* Samples taken of their skin, urine, and maybe stool and spinal fluid.
* Photos taken of their whole body. They can wear underwear and cover their eyes.
* Brain MRI. They will lie on a table that slides in and out of a metal cylinder. The scanner makes loud knocking noises so they can wear earplugs.
* Abdomen ultrasound. Sound waves take images of the body from the outside.
* Hand/wrist X-rays for young patients. They may have a full-body X-ray.
* DEXA bone density scan. Participants will lie on a table under a scanner.
* Echocardiogram and electrocardiogram for heart activity. Pads are stuck on the skin and the electrical activity of the heart is recorded.
* Tests of hearing, thinking, motor skills, and speech.
* Children participants may have tests done under sedation if it will benefit them directly.
* CDG participants may have other procedures during their visit. They may have follow-up visits every year.

DETAILED DESCRIPTION:
Study Description:

In this protocol, we propose to characterize the etiology and natural history of known, suspected or secondary CDGs to expand our knowledge about these disorders and provide access to patients of interest for research, teaching, and clinical experience.

Objectives:

The overall aim of this protocol is to advance our knowledge of primary, new, and secondary congenital disorders of glycosylation.

Study Population:

Participants 1 month or older will have been or will be referred to this protocol with a known or suspected CDG though only participants older than 2 years old will be evaluated as inpatients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants 1 month or older will have been or will be referred to this protocol with a known or suspected CDG. Participants over two years of age will be admitted only if they are medically stable and require admission to the Clinical Center for diagnosis. One or more probands may be admitted to the NIH Clinical Center for investigation as well as carrier family members.

Some participants will be relatives of patients with known CDG s, and their specimens will be obtained for the purpose of heterozygote testing and to serve as controls to help diagnose the proband. Participants may be seen as inpatients, outpatients or via Telehealth. In some cases, biologic samples may be obtained remotely and sent to the Gahl lab.

EXCLUSION CRITERIA:

* Participants under 1 month of age will not be seen at the NIH Clinical center because care is more readily proffered to older individuals at the Clinical Center.
* Participants over two years of age will not be admitted if they are medically unstable and do not require admission to the Clinical Center for diagnosis.
* Pregnant women and newborns are excluded.

Ages: 1 Month to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone with a congenital disorder of glycosylation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-03-07 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Expertise Establishment | Ongoing
  DescriptionTo employ consultations, physical examinations, and medical and genetic histories to establish expertise in these disorders appropriate to advise patients and physicians concerning diagnosis, prognosis, and therapy of CDGs.

SECONDARY OUTCOMES:
Secondary | Ongoing
  To use this protocol to recruit patients for potential future therapeutic studies.-To inspire the initiation of new, treatment-specific protocols.-To allow for collection of data on carrier family members enrolled in this protocol.-To perform standard genetic and non-genetic testing as indicated to identify new CDG s that may yield information about new variant(s) or cell biology.-To provide teaching and research cases for the NHGRI intramural community.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne A Wolfe, C.R.N.P., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
pending

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-HG-0071.html